CLINICAL TRIAL: NCT05530629
Title: Effect of Different Intensity Resistance Training on Energy Intake and Appetite Regulation Among Overweight and Obese College Girl
Brief Title: Effect of Resistance Training on Energy Intake and Appetite Regulation, 12-weeks Resistance Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Wang Qiang, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Wang Qiang
Record Dates: First submitted 2022-08-28; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Overweight; Obese
Keywords: Resistance training; Energy intake; Appetite; College Girl
MeSH Terms: conditions — Overweight; Obesity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: In this experiment, the three experimental groups will conduct different intensities resistance training, and the control group take the normal P.E. course.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity of resistance training (Experimental): The intensity of 75-80% 1RM is used for high intensity resistance training group. The number of repetitions of each set is relatively few, only 6-8 times. The rest time between sets is relatively long, 2-3 minutes, so that the participants can better adapt to this intensity.
  chest press, lat pull down, shoulder press and square, which are all trained through the multi-functional Smith machine.
  Bicep curl and triceps extension are operated by purchasing dumbbells with different weights.
  Leg extension and Leg curl use leg extension and curl machine Abdominal crunches and lower back exercises just do it by body weight training in yoga mat with abdominal curl and Lower back bridge
  Interventions: Device: resistance training
- Moderate intensity of resistance training (Experimental): The intensity of 60-65% 1RM is used for moderate intensity resistance training group. The repetition times of each set are relatively moderate, 10-12 times. The rest time between sets is relatively moderate, 1-2 minutes. The relative exercise volume of this group was consistent with that of other experimental groups chest press, lat pull down, shoulder press and square, which are all trained through the multi-functional Smith machine.
  Bicep curl and triceps extension are operated by purchasing dumbbells with different weights.
  Leg extension and Leg curl use leg extension and curl machine Abdominal crunches and lower back exercises just do it by body weight training in yoga mat with abdominal curl and Lower back bridge
  Interventions: Device: resistance training
- Low intensity of resistance training (Experimental): The intensity of 40-45% 1RM is used for low intensity resistance training group. The repetition times of each set are relatively more, 16-18 times. The rest time between groups is short, only about 1 minute, so that the participants can still maintain sufficient total exercise load under low intensity.
  chest press, lat pull down, shoulder press and square, which are all trained through the multi-functional Smith machine.
  Bicep curl and triceps extension are operated by purchasing dumbbells with different weights.
  Leg extension and Leg curl use leg extension and curl machine Abdominal crunches and lower back exercises just do it by body weight training in yoga mat with abdominal curl and Lower back bridge
  Interventions: Device: resistance training
- Normal P.E. course (Other): Carry out general teaching content according to the college syllabus.
  Interventions: Device: Normal P.E. course

INTERVENTIONS:
Device: resistance training — resistance training lasts for 12 weeks, three times a week, one hour each time, and the program of resistance training in the experimental group was divided into 10 exercises: Chest press, Lat pull down, Shoulder press, Squat, Leg extension, Leg curl, Bicep curl, Triceps extension, abdominal crunches, lower back exercises.
  Arms: High intensity of resistance training; Low intensity of resistance training; Moderate intensity of resistance training
Device: Normal P.E. course — Carry out general teaching content according to the college syllabus lasts for 12 weeks , three times a week, one hour each time, and the program of Normal P.E. course in the control group will be Physical recovery exercises, learn and practice queue formation, calisthenics, five step fists, long fist and Basic movements of Gymnastics gradually changed by week.
  Arms: Normal P.E. course

SUMMARY:
Resistance training is a common way of daily exercise which has a remarkable function in healthcare. It has been used in many diseases as a complementary method. Overweight and obesity are the sixth highest risk of death worldwide. In recent years, the data show that the rate of overweight obese among college students shows a significant increasing trend. The common characteristics of overweight and obese people are strong appetite which is difficult to be controled and sedentary. resistance training is a solid supplement to physical education and how to reduce appetite of overweight and obese college female students through resistance training is the key to increase their health by university sport course. The training plan divides the training intensity into three levels including 45-50% one repetition maximum(1RM), 60-65% 1RM, 45-50% 1RM, respectively plus control group. Therefore, this experimental research examines the effectiveness and the differences of three Intensities resistance training on energy intake and appetite regulation among overweight and obese college girl. Finally, to evaluate whether the resistance training can reduce the overweight and obese female college students' energy intake and appetite regulation

DETAILED DESCRIPTION:
On the basis of consulting relevant literature, this paper designs a 12 week teaching plan of resistance training through experimental design and quantitative research methods, combined with the characteristics of resistance training and the physiological characteristics of obese or overweight people. The purpose of this experiment is to provide a theoretical basis for improving the teaching methods of College Students' physical education, so as to improve the energy intake and appetite regulation of obese and overweight female college students, and then reduce their weight. And compared with ordinary daily physical education courses. Among them, the experimental group was divided into three groups, and the resistance training with intensity of 45-50% 1RM, 60-65% 1RM and 80-85% 1RM was carried out respectively. The control group carried out daily physical education teaching content. The number of participating samples in each group is 18 overweight or obese female college students, and the samples in each group are located in different campuses.

The first section of the training program of the experimental groups are warm up (10 mins) which including two parts. The first part is jogging and running indoor or stationary cycling outdoor with low intensity (5 minutes), the second part is muscle stretching: the Chinese eight set of radio kinetics (each movement 8 times) including stretch exercise, check augmentation exercise, kicking exercise, body side exercise, body rotation exercise, whole body exercise, jump exercise, cooling down exercise Then, the main resistance training section of the experimental group includes test press, late pull down, shoulder press, square, leg extension, leg curl, bicep curl, triceps extension, dominant crunches, lower back exercises In the last cool down phase, repeat the same content of muscle stretching as in the first part again.

Three times a week, with an interval of more than 48 hours. Each exercise of main resistance training takes 2 sets, and the repetition times of low intensity, medium intensity and high intensity are 16-18 times, 10-12 times and 6-8 times respectively. The rest time between low-intensity, medium-intensity and high-intensity groups is 1 minute, 1-2 minutes and 2-3 minutes respectively. The total duration of each training is about 1 hour, including warm up for about 10 minutes, main training time for about 45 minutes, and final cool down for about 5 minutes. In addition, the maximum strength was retested once at week 1, 5 and 9 respectively The control group only changed the resistance training part to normal P.E. course which carried out general teaching content according to the college syllabus, other settings are the same.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight or obese (BMI> 25)
2. Female
3. College students
4. Healthy

Exclusion Criteria:

1. The subjects lack regular and active exercise program in last three months
2. The subjects are not on a diet in last three months. c, Do not have regular menstrual cycle or approaching the normal menstrual cycle

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline BMI at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Obesity Degree.
Change from baseline body fat percentage at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Obesity Degree.
Change from baseline waist circumference at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Obesity Degree.
Change from baseline energy intake at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter will be recorded by Quantitative Daily Dietary Intake (QDI): three multiple-pass 24-hr recalls collected at each assessment time point by a research dietitian/technician. Analysis by Food Processor Nutrition Analysis Software (Version 9.6, 2005, ESHA Research, Salem, OR): recalls are analysed for calorie and macronutrient content
Change from baseline hunger at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter will be test by 100-mm visual analogue scale (VAS): test at 6:00-8:00 am following a 10h overnight fast, rate perceive appetite firstly. Then provide with a standardised caloric stimulus, at 30, 60, 90 and 120min post consumption rate perceived appetite again (r = 0.42 - 0.85).
  At every time point, both lengths of VAS 100 mm were used to record desire to eat, hunger, fullness, and prospective food consumption. The four standardized questions were:
  (i) how strong is your desire to eat? ("very weak" to "very strong"), (ii) how hungry do you feel? ("not hungry at all" to "as hungry as I've ever felt"), (iii) how full do you feel? ("not full at all" to "very full"), and (iv) how much food do you think you can eat? (Prospective food consumption; "nothing at all" to "a large amount") .
Change from baseline fullness at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter will be test by 100-mm visual analogue scale (VAS): test at 6:00-8:00 am following a 10h overnight fast, rate perceive appetite firstly. Then provide with a standardised caloric stimulus, at 30, 60, 90 and 120min post consumption rate perceived appetite again (r = 0.42 - 0.85).
  At every time point, both lengths of VAS 100 mm were used to record desire to eat, hunger, fullness, and prospective food consumption. The four standardized questions were:
  (i) how strong is your desire to eat? ("very weak" to "very strong"), (ii) how hungry do you feel? ("not hungry at all" to "as hungry as I've ever felt"), (iii) how full do you feel? ("not full at all" to "very full"), and (iv) how much food do you think you can eat? (Prospective food consumption; "nothing at all" to "a large amount") .
Change from baseline desire to eat at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter will be test by 100-mm visual analogue scale (VAS): test at 6:00-8:00 am following a 10h overnight fast, rate perceive appetite firstly. Then provide with a standardised caloric stimulus, at 30, 60, 90 and 120min post consumption rate perceived appetite again (r = 0.42 - 0.85).
  At every time point, both lengths of VAS 100 mm were used to record desire to eat, hunger, fullness, and prospective food consumption. The four standardized questions were:
  (i) how strong is your desire to eat? ("very weak" to "very strong"), (ii) how hungry do you feel? ("not hungry at all" to "as hungry as I've ever felt"), (iii) how full do you feel? ("not full at all" to "very full"), and (iv) how much food do you think you can eat? (Prospective food consumption; "nothing at all" to "a large amount") .
Change from baseline prospective food consumption at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter will be test by 100-mm visual analogue scale (VAS): test at 6:00-8:00 am following a 10h overnight fast, rate perceive appetite firstly. Then provide with a standardised caloric stimulus, at 30, 60, 90 and 120min post consumption rate perceived appetite again (r = 0.42 - 0.85).
  At every time point, both lengths of VAS 100 mm were used to record desire to eat, hunger, fullness, and prospective food consumption. The four standardized questions were:
  (i) how strong is your desire to eat? ("very weak" to "very strong"), (ii) how hungry do you feel? ("not hungry at all" to "as hungry as I've ever felt"), (iii) how full do you feel? ("not full at all" to "very full"), and (iv) how much food do you think you can eat? (Prospective food consumption; "nothing at all" to "a large amount") .
Change from baseline glucose at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Blood is collected into Vacutainers (BectonDickinson, Franklin Lakes, NJ) containing SST Gel (Becton Dickinson), Ethylenediaminetetraacetic acid(EDTA), or heparin and is immediately placed on ice and centrifuged (4 C, 1500g, 15 min). The serum or plasma obtained is stored in multiple aliquots at 75 C until assayed (in duplicate).
  Glucose is determined by the glucose oxidase method (Sigma-Aldrich Corp; 3.8% and 4.9% inter- and intraassay coefficients of variation) (70～140mg/dl or 3.9～7.8mmol/l)
Change from baseline leptin at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Blood is collected into Vacutainers (BectonDickinson, Franklin Lakes, NJ) containing Serum-separating tube(SST) Gel (Becton Dickinson), EDTA, or heparin and is immediately placed on ice and centrifuged (4 C, 1500g, 15 min). The serum or plasma obtained is stored in multiple aliquots at 75 C until assayed (in duplicate).
  Serum leptin is determined by an ELISA with a commercially available kit (EIA-2395, DRG, Marburg, Germany; 5.9% intraassay precision; 6.8% interassay accuracy; sensitivity of 0.5ng/ml).
Change from baseline adiponectin at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Blood is collected into Vacutainers (BectonDickinson, Franklin Lakes, NJ) containing SST Gel (Becton Dickinson), EDTA, or heparin and is immediately placed on ice and centrifuged (4 C, 1500g, 15 min). The serum or plasma obtained is stored in multiple aliquots at 75 C until assayed (in duplicate).
  Plasma adiponectin is analysed with a commercially available radioimmunoassay (RIA) (Linco Research, Inc., St. Charles, mo; 6.9% intraassay precision; 7.8% interassay accuracy; sensitivity of 0.5ng/ml.) (3~30μg/mL).
Change from baseline NPY at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Blood is collected into Vacutainers (BectonDickinson, Franklin Lakes, NJ) containing SST Gel (Becton Dickinson), EDTA, or heparin and is immediately placed on ice and centrifuged (4 C, 1500g, 15 min). The serum or plasma obtained is stored in multiple aliquots at 75 C until assayed (in duplicate).
  Neuropeptide Y is measured by Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) (NPY; Phoenix Europe Gesellschaft mit beschränkter Haftung (GmbH), Karlsruhe, Germany; Sensitivity of 0.13 ng/ml; Intra-assay variability <5%) (51.23～209.65 pg/ml).
Change from baseline Insulin at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Blood is collected into Vacutainers (BectonDickinson, Franklin Lakes, NJ) containing SST Gel (Becton Dickinson), EDTA, or heparin and is immediately placed on ice and centrifuged (4 C, 1500g, 15 min). The serum or plasma obtained is stored in multiple aliquots at 75 C until assayed (in duplicate).
  Insulin is measured with an immunoassay (Access Immunoassay System, Beckman Coulter, Fullerton, California (CA); 4.9% intraassay precision; 3.8% interassay accuracy; sensitivity of 0.5 μu/ml) (60-100mg/dl).
Change from baseline meal-time at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter record by Quantitative Daily Dietary Intake (QDI): three multiple-pass 24-hr recalls collected at each assessment time point by a research dietitian/technician. Analysis by Food Processor Nutrition Analysis Software (Version 9.6, 2005, ESHA Research, Salem, OR): recalls are analysed for the percentage of day and night total kcals intake separately.
Change from baseline stress of eating at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter measured by The Salzburg Stress Eating Scale (SSES) which is the first to specifically address the relationship of stress experiences and coping failure on the one hand and increases or decreases in food intake on the other hand. Higher SSES scores indicate eating more when stressed, while lower scores indicate eating less when stressed.
Change from baseline physical activity level at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter measured by Global Physical Activity Questionnaire (GPAQ). The GPAQ covers several components of physical activity, such as intensity, duration, and frequency, and it assesses three domains in which physical activity is performed (occupational physical activity, transport-related physical activity, and physical activity during discretionary or leisure time) comprising 16 questions (P1-P16). Since it was developed by World Health Organization (WHO) in 2002, the GPAQ has undergone a research program which shows that it is valid and reliable. It has become the most common tool in diagnostic and evaluation studies of physical activity globally.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, Doctor, Principal Investigator — University Putra Malaysia
Locations (1):
- YiChun Education College, Yichun, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
Because this is my doctoral thesis and it has certain confidentiality, I won't share it until I finish my doctoral thesis

REFERENCES:
- [Result] Bales CW, Hawk VH, Granville EO, Rose SB, Shields T, Bateman L, Willis L, Piner LW, Slentz CA, Houmard JA, Gallup D, Samsa GP, Kraus WE. Aerobic and resistance training effects on energy intake: the STRRIDE-AT/RT study. Med Sci Sports Exerc. 2012 Oct;44(10):2033-9. doi: 10.1249/MSS.0b013e318259479a. PMID 22525775
- [Derived] Wang Q, Xiao WS, Danaee M, Geok SK, Gan WY, Zhu WL, Mai YQ. Impact of resistance training intensity on body composition and nutritional intake among college women with overweight and obesity: a cluster randomized controlled trial. Front Public Health. 2025 May 30;13:1589036. doi: 10.3389/fpubh.2025.1589036. eCollection 2025. PMID 40520279
- See also: Description This article is from National Library of Medinice — http://pubmed.ncbi.nlm.nih.gov/22525775/